CLINICAL TRIAL: NCT03335124
Title: A Randomized, Double Blind, Placebo-Controlled Study to Investigate the Effects of Vitamin C, Hydrocortisone and Thiamine on the Outcome of Patients With Severe Sepsis and Septic Shock
Brief Title: The Effect of Vitamin C, Thiamine and Hydrocortisone on Clinical Course and Outcome in Patients With Severe Sepsis and Septic Shock
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to insufficient recruitment
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Sebastian Stefanovic, MD, Doctor of Medicine, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSEPSIS
Record Dates: First submitted 2017-10-25; First posted 2017-11-07 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Sepsis; Septic Shock; Critical Illness; Fluid Overload
Keywords: Sepsis; Vitamin C; Hydrocortisone; Thiamine; Critical Illness; Fluid Responsiveness; Hemodynamics
MeSH Terms: conditions — Sepsis; Shock, Septic; Critical Illness; Edema | interventions — Ascorbic Acid; Hydrocortisone; Adrenal Cortex Hormones; Thiamine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active substances (Experimental): Vitamin C: Vitamin C will be mixed as 1500 mg vitamin C in 50ml container, which will then be infused over 30 minutes to 1 hour. The bag will be labeled by the pharmacy as Vitamin C. The dosing schedule is 1500mg every 6 hours for 4 days or until discharge from the ICU.
  Hydrocortisone: Hydrocortisone will be mixed as 50 mg of Hydrocortisone in 50 ml of 0.9 % Sodium Chloride. Patients will be treated with hydrocortisone 50mg IV q 6 hourly for 4 days or until ICU discharge.
  Thiamine: Intravenous thiamine will be given in a dose of 200mg q 12 hourly for 4 days or until ICU discharge.
  Interventions: Drug: Vitamin C; Drug: Hydrocortisone; Drug: Thiamine
- Control (Placebo Comparator): Vitamin C placebo will consist of an identical container of 50cc normal saline (0.9% Sodium Chloride Injection) (but with no vitamin C) and will be labelled vitamin C. Placebo will be infused over 30-60 minutes as per the infusion instructions of the active vitamin. Hydrocortisone placebo will be provided in an identical 50 ml bag of 0.9% Sodium Chloride Injection. Placebo patients will receive a matching vial of 0.9% Sodium Chloride Injection.
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: Vitamin C — Vitamin C: Vitamin C will be applied as per instructions described in arm/group descriptions.
  Other Names: Ascorbic Acid
  Arms: Active substances
Drug: Hydrocortisone — Hydrocortisone: Hydrocortisone will be applied as per instructions described in arm/group descriptions.
  Other Names: Corticosteroids
  Arms: Active substances
Drug: Thiamine — Intravenous thiamine will be applied as per instructions described in arm/group descriptions.
  Other Names: B1 Vitamin
  Arms: Active substances
Drug: 0.9% Sodium Chloride Injection — 0.9 % Sodium Chloride will be applied as placebo as per instructions described in arm/group descriptions.
  Other Names: Normal Saline
  Arms: Control

SUMMARY:
The global burden of sepsis is substantial with an estimated 15 to 19 million cases per year; the vast majority of these cases occur in low income countries. New therapeutic approaches to sepsis are desperately required; considering the global burden of sepsis these interventions should be effective, cheap, safe and readily available. The aim is to study the synergistic effect of vitamin C, hydrocortisone and thiamine on survival in patients with severe sepsis and septic shock.

DETAILED DESCRIPTION:
AIM OF THE STUDY:

The goal is to determine the effects on clinical course and outcome of patients with severe sepsis and septic shock treated with vitamin C, hydrocortisone and thiamine.

BACKGROUND:

This study will be conducted in the intensive care unit of Department of Gastroenterology, University Medical Center (UMC) Ljubljana. All of the patients with severe sepsis and septic shock admitted to the Intensive Care Unit (ICU) in the past 12 hours will be screened for possible inclusion in the study. The diagnosis of severe sepsis and septic shock will be based on the 1992 American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference definitions.

PLAN OF THE STUDY:

After determining the eligibility for inclusion in our study, the investigators will acquire the written consent from the patient or relatives. The investigators (doctor on call) will randomize the patient either in the treatment or placebo group. The randomization will be done before-hand with the online tool Research Randomizer. After acquiring the randomized numbers, they will be placed in sealed envelopes. These envelopes will be available to the on-call doctor. The envelopes will then be sent to our outpatient clinic, where the studied substances will be mixed by a nurse, that will have no contact with the patients or the ICU staff. The substances will be marked with Vitamin C, Thiamine and Hydrocortisone, regardless if normal saline or the actual substances are inside the vials. Only this nurse will have the data regarding the contents of the vials.

Based on literature the investigators expect that survival and clinical course in sepsis and septic shock is correlated with fluid resuscitation and vasopressor use. Because of this, all of the included patients will be monitored with invasive hemodynamic monitoring (All of the patients will be monitored with the Edwards EV 1000 monitors).

All of the patients will be treated the same as per internationally recognized guidelines for treatment of septic shock. While the use of corticosteroids in severe sepsis is off-label, the patients will be informed of possible side-effects. This fact will also be written in the consent.

Neither the patients or the relatives will receive no financial compensation for study inclusion. During the hospitalization, the patients will receive three different substances in dosages, that are non toxic. During the study, there will be intermittent statistical analysis, and if increased mortality or severe side effects will be found then the study will be terminated. The confidentiality of personal data will be protected accordingly with the rules and laws of patient's privacy. The identity of patients will not be disclosed. The data acquired during the study will be available to the study participant. The anticipated costs will be covered by the Department of Gastroenterology, UMC Ljubljana. No financial compensation will be given to researchers.

During the study the following data will be acquired from the patients:

1. Age,
2. Sex,
3. Body weight,
4. Admitting diagnosis and source of infection,
5. Isolated pathogens,
6. Comorbidities,
7. The need for mechanical ventilation,
8. The use of vasopressors (all doses will be converted to Norepinephrine equivalents),
9. The duration of vasoactive therapy,
10. Daily urine output,
11. Fluid balance after 24 and 72 hours,
12. The presence of acute kidney failure
13. Duration of ICU stay and hospital stay,
14. Survival in ICU, hospital, after 28 and 60 days
15. Routine blood test for the first 4 days, a. creatinine b. White Blood Cells (WBC) c. Platelets d. Bilirubin e. Partial Pressure of Oxygen in Arterial Blood/Fraction of Inspired Oxygen (PaO2/FiO2) ratio e. procalcitonin (PCT) and procalcitonin clearance f. lactate g. blood samples will be stored for possible additional analysis

The patients' admission Acute Physiology and Chronic Health Evaluation (APACHE) II and APACHE IV scores will be recorded. The APACHE IV score allows calculation of the predicted hospital mortality and predicted ICU length of stay (LOS). The daily Sepsis-related Organ Failure Assessment (SOFA) score will be recorded for the first 4 treatment days.

Data analysis:

Summary statistics will be used to describe the clinical data and presented as mean ± standard deviation (SD), median with interquartile range (IQR) or percentages as appropriate. Chi squared analysis with Fisher's exact test (when appropriate) and Student's t test (Mann Whitney U test for non-normal distributions) were used to compare data between the active treatment group and the placebo group with statistical significance declared for probability values of 0.05 or less.

Data Safety & storage:

The main risk to subjects is the accidental release of Protected Health Information (PHI). Careful record management methods will be in place to ensure this type of privacy breach does not occur. The data set will be kept in a password-protected file and stored separately from the subject identification (ID) key in the locked office of the principal investigator. Only the research team will have access to this information, and will not disclose this information to any other person or entity. Three years after the completion of the study, all collected data will be destroyed by permanently deleting electronic copies.

EXPECTED RESULTS:

The investigators expect a faster recovery, shorter hospitalization, shorter use of vasoactive drugs and better survival in treatment group versus (vs.) control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe sepsis or septic shock within 12 hours of admission in our Intensive Care Unit (ICU).
* Informed consent.

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Do Not Resuscitate (DNR/DNI) with limitations of care
* Patients with fatal underlying disease who are unlikely to survive to hospital discharge (e.g.: disseminated malignant disease)
* Patients primarily admitted for acute coronary syndromes, acute cerebrovascular incidents or active gastrointestinal (GI) bleeds
* Patients that need immediate surgical treatment
* Patients with HIV and a cell count of cluster of differentiation 4 (CD4) cells < 50 mm2,
* Patients with known glucose-6 phosphate dehydrogenase (G-6PD) deficiency.
* Patients with severe sepsis/septic shock transferred from another hospital
* Patients with features of sepsis/septic shock > 24 hours
* Patients who require treatment with corticosteroids for an indication other than sepsis (chronic corticosteroid use, known Addison's Disease, Ulcerative colitis, Crohn's disease...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | From date of randomization till time of discharge, assessed up to 12 months
  We will compare mortality between the treatment and placebo groups during the hospitalization

SECONDARY OUTCOMES:
60 day mortality | 60 days from inclusion in the study
  We will compare mortality between the treatment and placebo groups after 60 days after inclusion in the study
28 day mortality | 28 days from inclusion in the study
  We will compare mortality between the treatment and placebo groups after 28 days after inclusion in the study
Time to vasopressor independence | Defined as the time from starting the active treatment/placebo to discontinuation of all pressors, till discharged from ICU, assessed in the first month
  Defined as the time from starting the active treatment/placebo to discontinuation of all pressors
PCT clearance | The first 4 days in Intensive Care Unit
  Clearance of calculated procalcitonin using the following formula: initial PCT minus PCT at 96 hours, divided by the initial PCT multiplied by 100.
Delta SOFA score | The first 4 days in Intensive Care Unit
  Delta Systemic Organ Failure Assesment score, defined as the initial SOFA score minus the day 4 SOFA score. The Sequential Organ Failure Assessment (SOFA) is a morbidity severity score and mortality estimation tool developed from a large sample of ICU patients throughout the world. The higher the value, the higher the mortality. The maximum score is 24, the lowest 0.
ICU length of stay (LOS) and ICU free days. | ICU free days is calculated as the number of days alive and out of the ICU to day 28
  ICU free days is calculated as the number of days alive and out of the ICU to day 28
Hospital Length of Stay | Hospital Length of Stay through the study completion, assessed up to 12 months
  The length of stay in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Stefanovic, MD, Principal Investigator — University Medical Center Ljubljana, Department of Gastroenterology
Locations (1):
- Department of Gastroenterology, UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For a year after the completion of the study
Access Criteria: Contributing authors that will sign the declaration of patient data confidentiality.

REFERENCES:
- [Background] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189
- [Background] Donnino MW, Andersen LW, Chase M, Berg KM, Tidswell M, Giberson T, Wolfe R, Moskowitz A, Smithline H, Ngo L, Cocchi MN; Center for Resuscitation Science Research Group. Randomized, Double-Blind, Placebo-Controlled Trial of Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. Crit Care Med. 2016 Feb;44(2):360-7. doi: 10.1097/CCM.0000000000001572. PMID 26771781
- [Background] Marik PE, Pastores SM, Annane D, Meduri GU, Sprung CL, Arlt W, Keh D, Briegel J, Beishuizen A, Dimopoulou I, Tsagarakis S, Singer M, Chrousos GP, Zaloga G, Bokhari F, Vogeser M; American College of Critical Care Medicine. Recommendations for the diagnosis and management of corticosteroid insufficiency in critically ill adult patients: consensus statements from an international task force by the American College of Critical Care Medicine. Crit Care Med. 2008 Jun;36(6):1937-49. doi: 10.1097/CCM.0b013e31817603ba. PMID 18496365
- [Background] Artenstein AW, Higgins TL, Opal SM. Sepsis and scientific revolutions. Crit Care Med. 2013 Dec;41(12):2770-2. doi: 10.1097/CCM.0b013e31829eb98f. PMID 23989175

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT03335124/Prot_SAP_000.pdf